CLINICAL TRIAL: NCT02988713
Title: Study to Characterize the Effects of Programming Spinal Cord Stimulation (SCS) in Patients Undergoing a Boston Scientific (BSC) SCS Temporary Trial
Brief Title: Study to Characterize Effects of Programming in SCS Patients Undergoing a Temporary Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 91153461
Record Dates: First submitted 2016-11-29; First posted 2016-12-09 (Estimated); Results first posted 2022-04-04 (Actual); Last update posted 2022-04-18 (Actual); Status verified 2022-04

CONDITIONS: Chronic Pain
Keywords: stimulation; chronic pain; back pain; leg pain
MeSH Terms: conditions — Chronic Pain; Back Pain

ARMS (1):
- Spinal cord stimulation (Experimental): Spinal cord stimulation (SCS) in patients undergoing a Boston Scientific (BSC) spinal cord stimulation (SCS) temporary trial
  Interventions: Device: Programming

INTERVENTIONS:
Device: Programming — Programming spinal cord stimulation (SCS) in patients undergoing a Boston Scientific (BSC) spinal cord stimulation (SCS) temporary trial

SUMMARY:
This is a prospective, multi-center, non-randomized, exploratory, single-arm study characterize the effects of programming spinal cord stimulation (SCS) in patients undergoing a Boston Scientific (BSC) spinal cord stimulation (SCS) temporary trial

ELIGIBILITY:
Key Inclusion Criteria:

* Study candidate is undergoing a spinal cord stimulation (SCS) trial of BSC neurostimulation system, per local directions for use (DFU).
* Subject signed a valid, Institutional Review Board (IRB)-approved informed consent form.
* Subject is 18 years of age or older when written informed consent is obtained.

Key Exclusion Criteria:

* Subject meets any contraindication in BSC neurostimulation system local directions for use (DFU).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2016-12-13 (Actual); Primary Completion 2020-12-02 (Actual); Study Completion 2020-12-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Roshini Jain, M.S., Study Director — Boston Scientific Corporation
Locations (2):
- United States (2):
  - Pacific Pain Management, Inc., Ventura, California
  - PCPMG Clinical Research Unit, LLC, Greenville, South Carolina

REFERENCES:
- [Derived] Zhu C, Esteller R, Block J, Lechleiter K, Frey R, Moffitt MA. Exploratory evaluation of spinal cord stimulation with dynamic pulse patterns: a promising approach to improve stimulation sensation, coverage of pain areas, and expected pain relief. Front Pain Res (Lausanne). 2024 Jan 31;4:1339892. doi: 10.3389/fpain.2023.1339892. eCollection 2023. PMID 38361978

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 35 subjects were enrolled in and started the study. 2 were withdrawn prior to the Programming Visit. 33 started the Programming Visit and 32 completed the study. Statistically relevant conclusions cannot be made from this small sample size.
Period: Overall Study
Arm/Group | Spinal Cord Stimulation
Started | 35
Completed | 32
Not Completed | 3
Not completed — Withdrawal by Subject | 1
Not completed — Subject's failure to meet study inclusion or exclusion criteria after enrollment | 2

BASELINE CHARACTERISTICS:
Arm/Group | Spinal Cord Stimulation
Number analyzed (Participants) | 35
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 18
  >=65 years | 17
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21
  Male | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 34
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 35
Work Status [Number; unit: participants] — Population: Analysis population n = 35. Measures are not mutually exclusive: one subject reported Work Status of both "Unemployed" and "Retired". Additionally, one subject did not report work status.
  participants
    Disability | 6
    Employed | 8
    Retired | 14
    Student | 1
    Unemployed | 6
    Not reported | 1

OUTCOME MEASURES:

1. Primary Outcome: Patient Comfort
Description: Number of participants reporting comfort level of stimulation sensation as "Very Comfortable" or "Slightly Comfortable"
Time Frame: An estimated average of 7 days post temporary trial procedure
Population: 32 subjects completing the Programming Visit
Measure: Count of Participants; unit: Participants
Arm/Group | Spinal Cord Stimulation
Number analyzed (Participants) | 32
Participants | 30

ADVERSE EVENTS:
Time Frame: Adverse events reported from enrollment to end of study (up to 15 days)
Arm/Group | Spinal Cord Stimulation
All-Cause Mortality (participants affected / at risk) | 0/35
Serious Adverse Events (participants affected / at risk) | 0/35
Other Adverse Events (participants affected / at risk) | 0/35

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-06-14): https://cdn.clinicaltrials.gov/large-docs/13/NCT02988713/Prot_SAP_000.pdf